CLINICAL TRIAL: NCT05721599
Title: Effectiveness of Integrated Care Combined Nutrition and Lifestyle Counselling in Frail Older Patients With Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB111-262-B
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Frailty; Diabetes; Lifestyle
Keywords: Frailty; Diabetes; Older adult; Integrated care; Nutrition; Lifestyle
MeSH Terms: conditions — Frailty; Diabetes Mellitus | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Structured integrated care model
  Interventions: Behavioral: Integrated care with nutrition and lifestyle counselling
- Control group (No Intervention): General outpatient care

INTERVENTIONS:
Behavioral: Integrated care with nutrition and lifestyle counselling — The structured care includes specialist care, integrated assessment, group health education, one-on-one nutrition and lifestyle guidance, online and face-to-face support group and case management.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of innovative integrated care in pre-frail or frail patients with diabetes over 65 years old. The main questions it aims to answer are:

* To establish innovative integrated care for frail elderly patients with diabetes combined with nutrition and lifestyle guidance.
* To evaluate the effectiveness of the intervention compared with general outpatient care.

Participants will receive 12 weeks of structured care including specialist care, integrated assessment, group health education, one-on-one nutrition and lifestyle guidance, online and face-to-face support group, and case management. Researchers will compare general outpatient care to see its effects on frailty, physical function, and blood sugar control.

DETAILED DESCRIPTION:
Frailty refers to a condition in which the body's reserves diminish with age, leading to a decreased ability to respond to stressors, making it difficult for individuals to maintain physiological stability and increasing susceptibility to diseases. The development of frailty often involves complex imbalances within the body's systems, such as the nervous system, endocrine system, immune system, and musculoskeletal system. Given the multifactorial nature of frailty, comprehensive assessments, and multifactorial interventions can improve functioning and reduce adverse outcomes in frail elderly individuals, including falls, hospitalization, or admission to nursing homes.

According to the American Diabetes Association guidelines, different A1c control targets can be established for elderly patients with diabetes based on their disease complexity, functionality, and cognitive status. Frailty, as a determinant of mortality in older adults, is also an important consideration in the treatment of diabetes. Furthermore, elderly patients with diabetes may experience a reduction in muscle strength and muscle mass, potentially leading to sarcopenia and subsequent frailty. Therefore, frailty and diabetes, two common health issues in the elderly, may mutually influence each other, altering the severity and treatment patterns of underlying diseases. Nutritional and lifestyle changes have the potential to slow down disability in frail elderly individuals with diabetes. While these recommendations are generally supported by guidelines, clinical evidence to support them is still needed. Past literature reviews have yet to conduct structured assessments of the effectiveness of nutritional and lifestyle guidance for frail elderly individuals with diabetes. Furthermore, in geriatric outpatient settings, a comprehensive integrated assessment should be used to establish treatment directions and plans for elderly patients with both frailty and diabetes, with ongoing monitoring.

In summary, aging is accompanied by disruptions in bodily systems, leading to the co-occurrence of frailty and diabetes, making them significant health issues during the aging process. Structured integrated care for frail elderly patients with diabetes, combining nutritional and lifestyle guidance, has the potential to reverse frailty, control blood sugar, and consequently delay disability. This study aims to investigate the effectiveness of innovative comprehensive assessments and care, including specialized care, integrated assessments, group health education, one-on-one nutritional and lifestyle guidance, online and face-to-face support group, and case management, on the improvement of frailty levels and blood sugar control in frail elderly patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* People aged 65 years or older.
* People with Clinical Frailty Scale: 4-7.
* People with a history of type II diabetes, use of diabetes medications, or HbA1c greater than or equal to 6.5%.
* People can understand the research process, meet the requirements of the research, and can sign the informed consent and participate in the following tracking.

Exclusion Criteria:

* People that are unable to cooperate with or accept intervention or follow-up.
* People with a history of type I diabetes.
* People use insulin injections or pumps.
* According to the PI's judgment, people with severe or poorly controlled conditions include acute diseases, severe infections, severe abnormal laboratory tests, or serious medical conditions with the following systems: cardiovascular, pulmonary, hepatic, nervous, mental, metabolic, renal, musculoskeletal, gastrointestinal, etc.
* People with severe visual or hearing impairment that prevent the completion of assessment and testing.
* People with malignant tumors that have just been diagnosed or are undergoing treatment or are still at risk of recurrence.
* People have received hormone therapy within three months before the trial or are expected to receive hormone therapy during the trial.
* People are currently or expected to join any other physical training courses or nutrition plans during the trial.
* Others are based on the judgment of the PI that participating in this trial may adversely affect the safety of the subjects, hinder the progress of the experiment, or interfere with the evaluation of the outcomes of the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline frailty | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Clinical Frailty Scale, max: 9, min: 1; higher score means worse outcome
Changes from baseline frail status | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Fatigue, Resistance, Ambulation, Illnesses, & Loss of Weight scale; max: 5, min: 0; higher score means worse outcome
Changes from baseline activities of daily living | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Barthel Index, max: 100, min: 0; higher score means better outcome
Changes from instrumental activities of daily living | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Instrumental Activities of Daily Living, max: 8, min: 0; higher score means better outcome
Changes from baseline cognition | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Mini-Mental Status Examination, max: 30, min: 0; higher score means better outcome
Changes from baseline depression | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Geriatric Depression Scale, max: 15, min 0; higher score means worse outcome
Changes from baseline nutritional status | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Mini-Nutritional Assessment-Short Form, max: 14, min: 0; higher score means better outcome
Changes from baseline fall risk assessment | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by fall risk assessment
Changes from baseline risk of sarcopenia | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by SARC-CalF, max: 20, min: 0; higher score means worse outcome
Changes from baseline physical activity | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by International Physical Activity Questionnaire
Changes from baseline quality of life | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Likert 7-point
Changes from baseline muscle strength measure by hand grip strength | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by hand grip strength
Changes from baseline walking speed | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by six-meter walking speed
Changes from baseline physical performance | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  measured by Short Physical Performance Battery
Change from baseline percentage of glycated hemoglobin (HbA1c) | baseline, 12 weeks, 24 weeks
  Change from baseline percentage of glycated hemoglobin (HbA1c)
Change from baseline concentration of low-density lipoprotein cholesterol (LDL-C) | baseline, 12 weeks, 24 weeks
  Change from baseline concentration of low-density lipoprotein cholesterol (LDL-C)
Change from baseline concentration of triglycerides | baseline, 12 weeks, 24 weeks
  Change from baseline concentration of triglycerides
Change from baseline concentration of high-density lipoprotein cholesterol (HDL-C) | baseline, 12 weeks, 24 weeks
  Change from baseline concentration of high-density lipoprotein cholesterol (HDL-C)
Change from baseline concentration of total cholesterol | baseline, 12 weeks, 24 weeks
  Change from baseline concentration of total cholesterol
Change from baseline body weight | baseline, 12 weeks, 24 weeks
  Change from baseline body weight
Change from baseline fat mass | baseline, 12 weeks, 24 weeks
  Change from baseline fat mass
Change from baseline muscle mass | baseline, 12 weeks, 24 weeks
  Change from baseline muscle mass
Change from baseline abdominal circumference | baseline, 12 weeks, 24 weeks
  Change from baseline abdominal circumference
Change from baseline calf circumference | baseline, 12 weeks, 24 weeks
  Change from baseline calf circumference

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Lun Kao, MD.PhD., Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No